CLINICAL TRIAL: NCT02349607
Title: A Double Blind, Double Dummy, Randomized, Placebo-controlled, 5 Period Cross-over Study To Examine The Effect Of Pf-05089771 Alone And In Combination With Pregabalin On Evoked Pain Endpoints In Healthy Volunteers Using Pregabalin And Ibuprofen As Positive Controls
Brief Title: Assessment of the Analgesic Effects of PF-05089771 and Pregabalin in Healthy Volunteers Using Evoked Pain Endpoints
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B3291010; 2014-004468-39 (EudraCT Number)
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
MeSH Terms: interventions — PF-05089771; Pregabalin; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- PF-05089771 300 mg (Experimental)
  Interventions: Drug: PF-05089771 300mg
- PF-05089771 300 mg + pregabalin 300 mg (Experimental)
  Interventions: Drug: PF-05089771 300 mg + pregabalin 300 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- pregabalin 300 mg (Active Comparator)
  Interventions: Drug: pregabalin 300 mg
- ibuprofen 600 mg (Active Comparator)
  Interventions: Drug: ibuprofen 600 mg

INTERVENTIONS:
Drug: PF-05089771 300mg — PF-05089771 300 mg
  Arms: PF-05089771 300 mg
Drug: PF-05089771 300 mg + pregabalin 300 mg — PF-05089771 300 mg + pregabalin 300 mg
  Arms: PF-05089771 300 mg + pregabalin 300 mg
Drug: Placebo — Placeco
  Arms: Placebo
Drug: pregabalin 300 mg — pregabalin 300 mg
  Arms: pregabalin 300 mg
Drug: ibuprofen 600 mg — ibuprofen 600 mg
  Arms: ibuprofen 600 mg

SUMMARY:
This study will examine the activity of PF-05089771 and pregabalin, alone and in combination on a panel of evoked pain tests carried out from 0.5 to 10 hours following oral dosing in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests. •Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs). •Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study. •Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing). •Any condition possibly affecting drug absorption (eg, gastrectomy). •A positive urine drug screen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Thermal pain detection threshold | 1-10 hours
Ultra-violet light sensitized pain detection threshold | 1-10 hours
Pressure pain tolerance threshold | 1-10 hours
Electrical pain tolerance threshold | 1-10 hours
Cold pressor tolerance threshold | 1-10 hours

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0.5-10
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0.5-10
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0.5-10
Electrical pain detection threshold | 0.5-10 hours
Electrical pain area under the visual analogue scale pain curve | 0.5-10 hours
Electrical pain post test visual analogue scale | 0.5-10 hours
Electrical pain post-cold pressor pain detection threshold | 0.5-10 hours
Electrical pain post cold pressor pain tolerance threshold | 0.5-10 hours
Electrical pain post cold pressor area under the visual analogue scale curve | 0.5-10 hours
Electrical pain post cold pressor post test visual analogue scale | 0.5-10 hours
Conditioned pain modulation response pain detection threshold | 0.5-10 hours
Conditioned pain modulation pain tolerance threshold | 0.5-10 hours
Conditioned pain modulation area under the visual analogue scale curve | 0.5-10 hours
Condition pain modulation post test VAS | 0.5-10 hours
Pressure pain detection threshold | 0.5-10 hours
Pressure pain area under the visual analogue scale curve | 0.5-10 hours
Pressure pain post test visual analogue scale | 0.5-10 hours
Cold pressor pain detection threshold | 0.5-10 hours
Cold pressor area under the visual analogue scale curve | 0.5-10 hours
Cold pressor post test visual analogue scale | 0.5-10 hours
PF-05089771 half life | 0.5-10 hours
Pregabalin half life | 0.5-10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Centre for Human Drug Research, Leiden, CL, Netherlands